CLINICAL TRIAL: NCT00298129
Title: Autonomic Imbalance and 24-h Blood Pressure Change in Patients With Chronic Renal Disease
Status: Completed | Type: Observational
Sponsor: Yokohama City University Medical Center (Other)
Other Study IDs: 7332-3
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2007-05-09 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus; Essential Hypertension; Renal Failure; Chronic Nephropathy
MeSH Terms: conditions — Diabetes Mellitus; Essential Hypertension; Renal Insufficiency | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring

SUMMARY:
Many patients with chronic renal disease show a loss of the nocturnal decline of blood pressure (non-dipper). However, the mechanism is not yet fully understood. We evaluate 24-hour blood pressure in patients with chronic renal disease using an ambulatory blood pressure monitoring device (A & D TM2425). We also analyze the power spectrum of heart rate variability as an index of autonomic cardiovascular modulation using the same device.

DETAILED DESCRIPTION:
The ratio of lower frequency (LF) and higher frequency (HF) heart rate rhythmic oscillations is expressed as an index of sympathovagal balance. Patients with chronic renal disease participate in the study. Blood pressure and power spectrum of heart rate variability for 24 hours are measured when they receive no medication for at least 1 week. The mean waking and sleeping time systolic and diastolic blood pressure are calculated. LF/HF ratios in the chronic renal disease are evaluated to calculate the waking/sleeping ratio for LF/HF.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with diabetes mellitus
* Hypertensive patients
* Hypertensive patients with renal disease
* Patients with chronic renal disease

Exclusion Criteria:

* Cardiac, hematologic or hepatic disease
* Cerebral infarction or hemorrhage
* Other major diseases.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2004-02; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gen Yasuda, MD, Principal Investigator — Yokohama City University Center Hospital
Locations (1):
- Yokohama City University Center Hospital, Yokohama, Japan

REFERENCES:
- [Background] Yasuda G, Nagasawa T, Umemura S, Shionoiri H, Ishii M. The impaired control of plasma renin activity in hypertensive patients with end-stage renal disease due to chronic glomerulonephritis. Clin Nephrol. 1994 Nov;42(5):300-8. PMID 7851031